CLINICAL TRIAL: NCT06633029
Title: Comparison of Patient Outcomes Between Retrospective Prismaflex HF20 Set and Historical Prospective Pediatric Continuous Renal Replacement Therapy (ppCRRT) Registry
Brief Title: Retrospective Analysis of Prismaflex HF20 Set Versus ppCRRT Registry
Status: Recruiting | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU602071
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Renal Failure (ARF); Acute Kidney Injury (AKI); Fluid Overload in Dialysis Patients
Keywords: Continuous Renal Replacement Therapy; CRRT
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Prismaflex HF20 cohort: Data collected from this study
  Pediatrics (weighing between 8 and 20 kg) who received CRRT with Prismaflex HF20 between 2008 to current in Canada or between 2020 to current in the US
  Interventions: Device: Prismaflex HF20
- Prismaflex M60 cohort: Data from ppCRRT registry used for comparison
  Pediatrics (weighing between 8 and 20 kg) who received CRRT with Prismaflex M60 sets
  Interventions: Device: Prismaflex M60

INTERVENTIONS:
Device: Prismaflex HF20 — CRRT fluid management and reduction of uremic toxins.
  Groups: Prismaflex HF20 cohort
Device: Prismaflex M60 — CRRT fluid management and reduction of uremic toxins.
  Groups: Prismaflex M60 cohort

SUMMARY:
A retrospective multicenter, observational design intended to capture data on pediatrics (weighing between 8 - 20 kg) who underwent continuous renal replacement therapy (CRRT) using the HF20 set. Data will be compared with a similar population (weighting 8-20 kg) from the ppCRRT registry who received CRRT with Prismaflex M60 sets.

DETAILED DESCRIPTION:
This study aims to compare patient outcomes after treatment with HF20 based CRRT to the historical ppCRRT registry. Data from eligible patient records will be collected, starting from January 2008 to most recent in Canada and from January 2020 to most recent in the US.

The ppCRRT registry used a prospective observational format whereby de-identified data on patients and CRRT circuits were collected from 13 participating centers across the US between 2001 JAN 01 and 2005 AUG 31. The registry's primary outcome measure was patient survival to ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patient weighed between 8 and 20 kg (17.6 - 44.1 lb).
2. Patient received medical care in an intensive care unit (ICU) and was treated with HF20 based CRRT.
3. Patient had a clinical diagnosis of AKI or ARF or fluid overload requiring CRRT.

Note: The cohort of patients treated with M60 sets from the ppCRRT registry (weighing 8 - 20 kg) are to meet inclusion criteria 1 and 3.

Exclusion Criteria:

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data from approximately 40 pediatric patients who had acute kidney injury (AKI), acute renal failure (ARF) or fluid overload requiring CRRT, weighed between 8 and 20 kg (17.6-44.1 lb), and were treated in the ICU with marketed HF20 based CRRT between 2008 to current in Canada or with HF20 product available under EUA between 2020 to current in the US, will be collected.
  Data will be compared with a similar population (weighing 8-20 kg) from the ppCRRT registry who received CRRT with Prismaflex M60 sets.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Survival to CRRT discontinuation | From CRRT initiation up to CRRT discontinuation of the first record of CRRT treatment with HF20/M60 (from January 2008 to present in Canada, and from January 2020 to present in the US)
  The proportion of patients who completed HF20/M60 based CRRT
Survival to ICU discharge | From ICU admission up to ICU discharge as related to of the first record of CRRT treatment with HF20/M60 (from January 2008 to present in Canada, and from January 2020 to present in the US)
  The proportion of patients who were released from the ICU

SECONDARY OUTCOMES:
ICU length of stay | From ICU admission up to ICU discharge as related to of the first record of CRRT treatment with HF20/M60 (from January 2008 to present in Canada, and from January 2020 to present in the US)
  The duration of time (in days) patients were in the ICU
CRRT duration | From CRRT initiation up to CRRT discontinuation of the first record of CRRT treatment with HF20/M60 (from January 2008 to present in Canada, and from January 2020 to present in the US)
  The duration of time (in days) HF20/M60 based CRRT was performed
AEs of relevance for HF20 | From CRRT initiation up to CRRT discontinuation of the first record of CRRT treatment with HF20 (from January 2008 to present in Canada, and from January 2020 to present in the US)
  AEs of relevance (non-serious and serious) documented in the patient's medical records that occurred during HF20 based CRRT treatment within the collection period (i.e., from 2008 to present for patients in Canada or 2020 to present for US patients).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Seattle Children's Hospital Research and Foundation, Seattle, Washington